CLINICAL TRIAL: NCT04560933
Title: A Prospective, Observational Study Evaluating Seroprevalence and Rate of Seroconversion of Antibodies Against Adeno-associated Virus (AAV) Serotypes and Exploratory Vectors in Subjects With Hemophilia A in the United States
Brief Title: A Study to Evaluate Seroprevalence and Seroconversion of Antibodies to Adeno-Associated Virus (AAV) in Patients With Hemophilia A
Acronym: SAAVY
Status: Completed | Type: Observational
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: 270-701
Record Dates: First submitted 2020-09-15; First posted 2020-09-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample collection for AAVx serotypes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Blood sample collection — Blood sample collection

SUMMARY:
To quantify the seroprevalence of antibodies to AAV5, AAV6, and AAV8 and the seroconversion rate over varying follow-up intervals in subjects with hemophilia A

DETAILED DESCRIPTION:
This is a single-center, decentralized, patient-centered, prospective, observational study utilizing biospecimen samples collected from hemophilia A subjects across the United States to evaluate and characterize seroprevalence and the rate of seroconversion of antibodies against AAV serotypes and exploratory vectors, and to investigate the associated factors that may influence the vector titers.

Relevant medical findings will also be collected from the subject, as well as symptoms related to hemophilia A. The collection of medical history may include major illnesses, diagnoses, and surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with Hemophilia A
* Subjects aged 18years or over at time of entry

Exclusion Criteria:

* Currently participating in an interventional study of any investigational product, device or procedure.
* Subjects who have been previously treated with AAV vector gene therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with Hemophilia A
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Assess the Seroprevalence of antibodies to AAV vectors in patients with hemophilia A | Baseline
  To assess the Seroprevalence of antibodies to AAV vectors in patients with hemophilia A at Baseline
Assess the rate of Seroconversion of antibodies to AAV vectors in patients with hemophilia A | Change from baseline through Week 12

SECONDARY OUTCOMES:
To describe and characterize AAV vector titer values in subjects with Hemophilia A | Change from baseline through Week 12
  To describe and characterize AAV vector titer values in subjects with Hemophilia A
To describe and characterize AAV vector titer values in subjects with Hemophilia A | Change from baseline through Week 24
  To describe and characterize AAV vector titer values in subjects with Hemophilia A

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Flach, MD, Principal Investigator — Covance
Locations (1):
- Covance Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No